CLINICAL TRIAL: NCT05356637
Title: Prospective Trial of Bipolar Sealer for Reduction of Intra-Operative Blood Loss in Total Hip Arthroplasty Utilizing the Anterior Hip Approach
Brief Title: Bipolar Sealer for Reduction of Blood Loss in Anterior Total Hip Arthroplasties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: North Texas Medical Research Institute, PLLC (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Mohammad Umar Burney, MD, Principal Investigator, Clinical Medical Director, North Texas Medical Research Institute, PLLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN-012022-01
Record Dates: First submitted 2022-03-28; First posted 2022-05-02 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Hip; Blood Loss
MeSH Terms: conditions — Osteoarthritis, Hip; Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention Group Receiving Fastseal (Other)
  Interventions: Device: Werewolf Fastseal 6.0

INTERVENTIONS:
Device: Werewolf Fastseal 6.0 — bi-polar hemostatic wand

SUMMARY:
The overall objectives and purpose of this study is to show that the Smith and Nephew Werewolf Fastseal 6.0 Bipolar Sealer is an effective tool to aide the surgical team in providing significant hemostasis during anterior total hip arthroplasty which would subsequently improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The patient is to undergo a standard of care primary total hip replacement for degenerative joint disease. All devices are to be used according to the approved indications, this includes the FDA approved Werewolf Fastseal Bipolar Device.
* The patient is expected to have an outpatient status and will be discharged <23 hours.
* Individuals who are able to speak, read, and comprehend the Institutional Review Board approved Informed Consent Document and willing and able to provide informed patient consent for participation in the study.
* Individuals who are willing and able to complete follow-up visits and questionnaires as specified by the study protocol.
* Individuals who are not bedridden per the discretion of the investigator (The intent of "not bedridden" means a permanent situation, not a temporary situation as in a hip fracture or trauma case).
* Individuals who are a minimum age of 21 years and less than 80 years at the time of consent.

Exclusion Criteria:

* Active local or systemic infection.
* Hematologic disease either inherited or acquired, that would predispose the patient to anemia or increased intra-operative blood loss
* Currently taking anti-coagulation medications more than 81 mg aspirin every day.
* Platelet disorder either inherited or acquired with a serum platelet level <150,000 platelets per microliter.
* Coagulopathy as seen with routine lab work
* Unstable/uncontrolled cardiovascular disease such as congestive heart failure, hypertension, or renal disease such as GFR <70, in the opinion of the investigative team and PI.
* Excessive alcohol intake or tobacco use, in the opinion of the investigator.
* Uncontrolled diabetes mellitus with hemoglobin a1c >7.5%.
* Established history of previous venous thrombotic events (VTE).
* Loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified.
* The subject is a woman who is pregnant or lactating.
* Subject had a contralateral amputation.
* Previous partial hip replacement in affected hip.
* Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three months.
* Contralateral hip was replaced less than 3 months prior to surgery date, contralateral hip is already enrolled in the study, or simultaneous or staged hip replacement is planned
* Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
* Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
* Subject, in the opinion of the Investigator, is a drug or alcohol abuser or has a physical or psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
post-operative hemoglobin | taken at 48-72 hours post op
  obtained from point of care testing (hemocue hgb 801 device) in clinic (g/dL)
intra-operative total blood loss | taken at time of surgery
  total blood loss approximated in milliliters from measuring output in suction canister and input from fluid bags with measurement markings

SECONDARY OUTCOMES:
Post-operative need for transfusion | 6 weeks post operative period
  measured in units given
Mean operative time ("skin to skin") | intra-operative
  measured in hh:mm:ss
incidence of VTE | for post-operative 6 weeks
  absolute value, diagnosed via VDS within 6 weeks
patient reported pain scoring | measured at preop, 2 weeks, 6 weeks
  numerical score, patient reported. ranges from 0 = no pain to 10 = worst pain
patient reported pain prescription drug usage | measured at post-operative period of 6 weeks
  patient reported as far as pain rx used and how many pills/hr (e.g. "I use norco 5-325. I pill every 8 hours currently").
Harris Hip Score analysis 6 weeks post operative visits | measured at preop, and at 6 weeks
  established orthopaedic score used to measure functionality of the hip, reported as numerical value. this will be aggregated and reported as a mean at study completion
length of hospital stay | post-operative for 6 weeks
  This will be measured with chart review and reported as "0" for <24 hour discharge and each subsequent 24 hour period as "1, 2, 3, etc".

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad U Burney, MD, Principal Investigator — NTMRI, OSD
Locations (2):
- United States (2):
  - Texas Health Sugery Center - Rockwall, Rockwall, Texas
  - Baylor Scott & White - Lake Pointe Medical Center, Rowlett, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gao FQ, Li ZJ, Zhang K, Sun W, Zhang H. Four Methods for Calculating Blood-loss after Total Knee Arthroplasty. Chin Med J (Engl). 2015 Nov 5;128(21):2856-60. doi: 10.4103/0366-6999.168041. PMID 26521781
- [Background] Nichols CI, Vose JG. Clinical Outcomes and Costs Within 90 Days of Primary or Revision Total Joint Arthroplasty. J Arthroplasty. 2016 Jul;31(7):1400-1406.e3. doi: 10.1016/j.arth.2016.01.022. Epub 2016 Jan 21. PMID 26880328
- [Background] Marulanda GA, Ulrich SD, Seyler TM, Delanois RE, Mont MA. Reductions in blood loss with a bipolar sealer in total hip arthroplasty. Expert Rev Med Devices. 2008 Mar;5(2):125-31. doi: 10.1586/17434440.5.2.125. PMID 18331175
- [Background] Procyk S. The Transcollation: Short Hospitals Stay and Accelerated Recovery in Total Hip and Knee Arthroplasties Using a Radiofrequency Bipolar Sealer - an Innovative Approach in the Conceptualization of the Surgical Gesture. Natl Acad of Surg 2015:15(2):87-97.
- [Background] Rosenberg AG. Reducing blood loss in total joint surgery with a saline-coupled bipolar sealing technology. J Arthroplasty. 2007 Jun;22(4 Suppl 1):82-5. doi: 10.1016/j.arth.2007.02.018. PMID 17570284
- [Result] Ackerman SJ, Tapia CI, Baik R, Pivec R, Mont MA. Use of a bipolar sealer in total hip arthroplasty: medical resource use and costs using a hospital administrative database. Orthopedics. 2014 May;37(5):e472-81. doi: 10.3928/01477447-20140430-59. PMID 24810825
- [Result] Bierbaum BE, Callaghan JJ, Galante JO, Rubash HE, Tooms RE, Welch RB. An analysis of blood management in patients having a total hip or knee arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):2-10. doi: 10.2106/00004623-199901000-00002. PMID 9973048